CLINICAL TRIAL: NCT04819724
Title: LiTrans - Influence of Additional Weight Carrying on Load-induced Changes in Glenohumeral Translation in Patients With Rotator Cuff Tear - a Translational Approach
Brief Title: Load-induced Changes in Glenohumeral Translation in Patients With Rotator Cuff Tear
Acronym: LiTrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-00182; mu21Muendermann
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tear
Keywords: glenohumeral translation; Load-induced Glenohumeral Translation (liTr ); Load-induced Muscle Activation (liMA)
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: cross-sectional experimental multimodal (clinical, biomechanical, radiological) data collection with multiple conditions and a control group
Masking Description: Blinding to the experimental condition is not possible because of the obvious differences between conditions (additional load). However, the person processing the data will be blinded to the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: patient group (unilateral rotator cuff tear) (Other): Group 1: 25 patients with unilateral symptomatic rotator cuff tear
  Interventions: Diagnostic Test: 3D motion analysis; Diagnostic Test: isometric shoulder strength by dynamometer; Diagnostic Test: fluoroscopic images of each shoulder; Diagnostic Test: Bilateral shoulder Magnetic Resonance Imaging (MRI); Other: data collection by health questionnaires
- Group 2: control group (asymptomatic volunteers) (Other): Group 2: (asymptomatic volunteers) 25 asymptomatic control subjects (age and sex distribution matching the patient group)
  Interventions: Diagnostic Test: 3D motion analysis; Diagnostic Test: isometric shoulder strength by dynamometer; Diagnostic Test: fluoroscopic images of each shoulder; Diagnostic Test: Bilateral shoulder Magnetic Resonance Imaging (MRI); Other: data collection by health questionnaires
- Group 2: young control group (young asymptomatic volunteers) (Other): Group 3: (young asymptomatic volunteers) 25 asymptomatic control subjects, 20 to 30 years (sex distribution matching the patient group)
  Interventions: Diagnostic Test: 3D motion analysis; Diagnostic Test: isometric shoulder strength by dynamometer; Diagnostic Test: fluoroscopic images of each shoulder; Diagnostic Test: Bilateral shoulder Magnetic Resonance Imaging (MRI); Other: data collection by health questionnaires

INTERVENTIONS:
Diagnostic Test: 3D motion analysis — 30° arm abduction in the scapular plane will be performed with and without a handheld weight of 1, 2, 3, and 4 kg. All movements will be done bilaterally. Electromyographic (EMG) data of arm and trunk muscles will be recorded using surface electrodes. Participants will be asked to perform full arm abduction with different rotations (internal, neutral and external rotation), flexion and internal-/external rotations movements (without additional handheld weight).
Diagnostic Test: isometric shoulder strength by dynamometer — isometric shoulder strength for abduction and internal/external rotation will be assessed with a isometric shoulder strength for abduction and internal/external rotation will be assessed with a dynamometer
Diagnostic Test: fluoroscopic images of each shoulder — fluoroscopic images (Multitom Rax, Siemens Healthineers, Erlangen, Germany) of each shoulder will be taken during the 30° arm abduction test with and without a handheld weight (0, 2, and 4kg)
Diagnostic Test: Bilateral shoulder Magnetic Resonance Imaging (MRI) — MRI of both shoulders will be taken
Other: data collection by health questionnaires — data collection by health questionnaires

SUMMARY:
The study is to investigate the dose-response relationship between load-induced muscle activation (liMA) and load-induced glenohumeral translation (liTr) in patients with rotator cuff tears and asymptomatic control subjects.

Furthermore the study is to investigate the in vivo dose-response relationship between additional weight and glenohumeral translation, to understand the biological variation in liTr, the influence of disease pathology on the liTr, the potential compensation by muscle activation and muscle size, and the influence of liTr on patient outcomes.

DETAILED DESCRIPTION:
This project is to test the overall hypothesis that rotator cuff tear affects glenohumeral translation and that this functional instability depends on additional load applied, on anatomical and morphological variations, and on type and severity of the injury. The study is to investigate the dose-response relationship between load-induced muscle activation (liMA) and load-induced glenohumeral translation (liTr) in patients with rotator cuff tears and asymptomatic control subjects.

Furthermore the study is to investigate the in vivo dose-response relationship between additional weight and glenohumeral translation, to understand the biological variation in liTr, the influence of disease pathology on the liTr, the potential compensation by muscle activation and muscle size, and the influence of liTr on patient outcomes.

This study entails cross-sectional experimental multimodal (clinical, biomechanical, radiological) data collection with multiple conditions and a control group.

ELIGIBILITY:
We will examine a cohort of 75 subjects:

* Group 1: 25 patients with unilateral symptomatic rotator cuff tear between 45 and 85 years
* Group 2: 25 asymptomatic control subjects (age and sex distribution matching the patient group) Group 3: 25 sex matched young asymptomatic control subjects between 20 and 30 years

Inclusion criteria patients:

* Diagnosed unilateral rotator cuff tear
* Partial or complete supraspinatus muscle tear
* With or without injury to other rotator cuff muscles

Exclusion criteria patients:

* Prior operative treatment of the ipsilateral shoulder or elbow
* Clinical history or symptoms of the contralateral glenohumeral joint
* Range of motion <30° in abduction and flexion

Inclusion criteria asymptomatic control subjects:

- No previous known elbow and shoulder injury or symptoms

Exclusion criteria asymptomatic control subjects:

* Clinical history of the glenohumeral joint
* Prior conservative or operative treatment of the shoulder or elbow
* Range of motion <90° in abduction and flexion

General exclusion criteria:

* Inability to provide informed consent
* Body mass index (BMI) > 35 kg/m2 (Excessive skin movement)
* Neuromuscular disorders affecting upper limb movement
* Additional pathologies that influence the mobility of the shoulder joints
* Contraindications for MRI (e.g. neurostimulator and claustrophobia)
* Prior neuromuscular impairment (e.g. stroke)
* Diagnosed active rheumatic disorder
* Other major medical problems
* Pregnancy
* Patients currently enrolled in another experimental (interventional) protocol

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Disabilities of arm, shoulder and hand (Quick DASH) questionnaire | at baseline (approximate duration for all questionnaires: 20 minutes)
  30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale (1 being no difficulty, 5 being unable).
Constant Score | at baseline (approximate duration for all questionnaires: 20 minutes)
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | at baseline (approximate duration for all questionnaires: 20 minutes)
  The American Shoulder and Elbow Surgeons Shoulder Score (ASES) is a mixed outcome reporting measure, applicable for use in all patients with shoulder pathology regardless of their specific diagnosis. The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain, instability, and activities of daily living. The pain and functional portions are summed to obtain the final ASES score with higher scores indicating better outcomes.
Subjective Shoulder Value (SSV) | at baseline (approximate duration for all questionnaires: 20 minutes)
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.
numerical pain rating scale (NRS) score | at baseline (approximate duration for all questionnaires: 20 minutes)
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults (from 0-10: "0" = no pain. "10" = the most intense pain imaginable)
Loaded shoulder abduction test with motion analysis | at baseline (approximate duration for motion analysis: 50 minutes)
  The subject will lift their arm to 30° shoulder abduction in the scapular plane, data will be captured holding 0, 1, 2, 3, and 4 kg, respectively, in their hand. Reflective surface markers will be placed bilaterally on the participants' trunk and arms. Position of these markers will be recorded using infrared cameras that only record the reflections of the markers. Additionally, inertial sensors will be positioned on the subjects' thorax, scapulae, humeri and forearms.
Loaded shoulder abduction test with single plane fluoroscopic images | at baseline (approximate duration for motion analysis: 50 minutes).
  fluoroscopic images (Multitom Rax, Siemens Healthineers, Erlangen, Germany) of each shoulder will be taken during the 30° arm abduction test with and without a handheld weight (0, 2, and 4kg)
Load-induced muscle activity from electromyography (EMG) | at baseline (approximate duration for motion analysis: 50 minutes)
  During arm movements in the loaded shoulder test and muscle strength tests, muscle activation of the infraspinatus, biceps brachii, anterior, middle and posterior part of the deltoid, clavicular part of the pectoralis major, latissimus dorsi and the upper part of the trapezius will be measured bilaterally using a 16-channel EMG system
Glenohumeral translation from single plane fluoroscopy | at baseline (approximate duration for motion analysis: 50 minutes)
  the vertical distance of the glenohumeral joint centre (GHJC) and the radiopaque acromion marker will be measured. Fluoroscopy (FL) based liTr will be calculated for each participant as the slope of the regression of the negative GHJC to acromion distance measurements on the load magnitude.
Glenohumeral translation from instrumented motion analysis | at baseline (approximate duration for motion analysis: 50 minutes)
  The vertical distance of the GHJC to the acromion marker will be calculated for a neutral trial and with the arm in 30° shoulder abduction for each loading condition. Motion analysis (MA) based liTr will be calculated for each participant as the slope of the regression of the negative GHJC to acromion distance measurements on the load magnitude
Critical shoulder angle (CSA) | at baseline (approximate duration for motion analysis: 50 minutes)
  Subject's CSA will be measured on an anterior-posterior double-obliquity fluoroscopy image of the shoulder as the angle subtended by a line parallel to the glenoid and a line through the inferior-lateral edge of the glenoid and the inferior-lateral edge of the acromion. The CSA is reproducible and significantly greater in patients with rotator cuff tears than the general population. High angles (>35°-38°) have been associated with rotator cuff tears and greater joint instability.
Glenoid inclination (GI) | at baseline (approximate duration for motion analysis: 50 minutes)
  GI will be measured on the fluoroscopy image as the angle between a line from the upper to the lower glenoid rim (glenoid plane) and a second line set on the floor of the supraspinous fossa. Abnormal GI might be associated with rotator cuff tears and superior humeral head migration.
Greater tuberosity angle (GTA) | at baseline (approximate duration for motion analysis: 50 minutes)
  GTA will be measured as the angle between a line parallel to the humerus diaphysis through the GHJC and a line from the upper border of the humeral head to the most superolateral edge of the greater tuberosity. A GTA of more than 70° has been observed to predict rotator cuff tear.
Muscle cross sectional area (MCSA) | at baseline (approximate duration is approximately 1 hour and 15 minutes)
  The MCSA of all rotator cuff muscles will be measured at two different positions on parasagittal reformatted images. MCSA of the deltoid will also be measured on the axial plane at the middle of the glenoid.
Tear size retrieved from MR images | at baseline (approximate duration is approximately 1 hour and 15 minutes)
  Tear size will be classified into partial (1) or complete supraspinatus muscle tear (2).
Tear type retrieved from MR images | at baseline (approximate duration is approximately 1 hour and 15 minutes)
  Tear type will be classified into supraspinatus tear without injury to other rotator cuff muscles (type A) and with injury to other rotator cuff muscles (type B). Both will be used as indicators for injury severity
Isometric shoulder muscle strength for abduction and internal/external rotation | at baseline (approximate duration: 40 minutes).
  Shoulder muscle strength will be tested under isometric conditions using a dynamometer. The maximum of 3 trials will be calculated and recorded as the participant's maximum isometric strength.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Mündermann, Prof. Dr., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Croci E, Hess H, Genter J, Baum C, Kovacs BK, Nuesch C, Baumgartner D, Gerber K, Muller AM, Mundermann A. Severity of rotator cuff disorders and additional load affect fluoroscopy-based shoulder kinematics during arm abduction. J Orthop Traumatol. 2024 Jun 8;25(1):30. doi: 10.1186/s10195-024-00774-2. PMID 38850466
- [Derived] Croci E, Warmuth F, Baum C, Kovacs BK, Nuesch C, Baumgartner D, Muller AM, Mundermann A. Load-induced increase in muscle activity during 30 degrees abduction in patients with rotator cuff tears and control subjects. J Orthop Traumatol. 2023 Aug 4;24(1):41. doi: 10.1186/s10195-023-00720-8. PMID 37542140
- [Derived] Croci E, Eckers F, Nuesch C, Aghlmandi S, Kovacs BK, Genter J, Baumgartner D, Muller AM, Mundermann A. Load-Induced Glenohumeral Translation After Rotator Cuff Tears: Protocol for an In Vivo Study. JMIR Res Protoc. 2022 Dec 23;11(12):e43769. doi: 10.2196/43769. PMID 36563028